CLINICAL TRIAL: NCT00521027
Title: A Prospective, Comparative, Single-centre Clinical Evaluation to Investigate the Skin-to-skin Time of the First Surgical Debridement of Lower Extremity Ulcers With VERSAJET™ Hydrosurgery System and Conventional Debridement Techniques.
Brief Title: Study Comparing VERSAJET With Conventional Surgical Procedures in the Removal of Unhealthy Tissue From Lower Limb Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE025VJT
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Diabetic Foot; Varicose Ulcer; Pressure Ulcer
Keywords: Debridement; hydrosurgery; Versajet; leg ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Other): Debridement with Versajet Hydrosurgery system
  Interventions: Device: Versajet Hydrosurgery System
- Control (Other): Conventional surgical debridement techniques
  Interventions: Procedure: Conventional surgical debridement techniques

INTERVENTIONS:
Device: Versajet Hydrosurgery System — Debridement with Versajet Hydrosurgery System
  Arms: Treatment
Procedure: Conventional surgical debridement techniques — Conventional surgical debridement with scalpel and pulse lavage
  Arms: Control

SUMMARY:
The purpose of this study is to compare the VERSAJET™ device with conventional surgical procedures (performed with a scalpel) in the debridement (removal of unhealthy tissue) of lower limb ulcers.

It is hypothesised that the time taken to debride lower limb ulcers will be quicker with the VERSAJET™ device than with conventional surgical procedures.

DETAILED DESCRIPTION:
This is prospective, comparative clinical evaluation to investigate whether there is a reduction in the skin-to-skin time of the first surgical debridement with VERSAJET™, compared to conventional debridement techniques. Skin-to-skin time is defined as the time of incision to the end time of debridement (wound ready for dressing application). Conventional debridement is defined as scalpel plus pulse lavage.

The purpose of this comparison is to demonstrate the resource savings which VERSAJET™ may provide in terms of operating room (OR) and personnel time, in addition to the potential to reduce the procedure, and possibly anaesthetic, time for the patient. It is envisaged that this information, combined with the costs associated with the procedure, will also provide valuable economic data to help justify the use of VERSAJET™ from a financial perspective and support the future commercial success of the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age.
* Males and females (provided they are not pregnant or, if of reproductive age, are using contraception).
* Patients with a venous stasis, diabetic foot or decubitus reference ulcer located between the tibia and foot.
* Patients undergoing surgical debridement of their reference ulcer in the operating room (OR).
* Patients undergoing their first surgical debridement of the reference ulcer.
* Patients suitable for debridement of their reference ulcer with both VERSAJET™ and conventional debridement techniques.
* Patients who are able to understand the evaluation and are willing and able to provide written consent to participate in the evaluation.

Exclusion Criteria:

* Patients with clinical signs of infection in the reference ulcer (e.g. purulence and / or odour).
* Patients with haemophilia
* Patients who have been treated with topical steroids, systemic immunosuppressants (including corticosteroids), anticoagulants or cytotoxic chemotherapy in the last 30 days, or who are anticipated to require such medications during the course of the study.
* Patients known to have Acquired Immunodeficiency Syndrome (AIDS) or known to be infected with Human Immunodeficiency Virus (HIV).
* Patients who suffer from acute or chronic bacterial, viral or fungal skin diseases that would interfere with wound healing.
* Patients with a known history of poor compliance with medical treatment.
* Patients who have participated in this evaluation previously or are currently participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-04; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Reduction in the average skin-to-skin time of the first surgical debridement with VERSAJET™, compared to conventional debridement techniques. | During surgery

SECONDARY OUTCOMES:
Difference in the total average time of the debridement procedure, including preparation, skin-to-skin and recovery, according to the debridement technique. | Entry into OR holding area to discharge from recovery room
Difference in outcomes of the procedure, according to the debridement technique in terms of; time to wound closure, number of subsequent debridements, number of serious adverse events | 3 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Wayne J Caputo, DPM, Principal Investigator — Clara Maass Medical Center
Locations (1):
- Clara Maass Medical Center, Belleville, New Jersey, United States